CLINICAL TRIAL: NCT02133729
Title: IMAGE (Metabolic Risk During Gestation) : Prospective Study of Women With Gestational Diabetes
Brief Title: Metabolic Risk Following Gestational Diabetes Mellitus
Acronym: IMAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2010.649
Record Dates: First submitted 2014-04-25; First posted 2014-05-08 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Blood Specimen Collection; Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gestational diabete (Experimental)
  Interventions: Other: Blood sampling and OGTT

INTERVENTIONS:
Other: Blood sampling and OGTT

SUMMARY:
Gestational diabetes (GDM) is defined by abnormal glucose tolerance during gestation. This complication occurs in 4-10% and is associated with fetal complications and macrosomia. In addition, women with GDM have an increased risk to develop type 2 diabetes after delivery. Despite recommendations, it is difficult to follow-up all women with GDM during the postpartum period due to high numbers of subjects that exceed usual healthcare resources. It is therefore necessary to focus clinical attention toward women at high risk of type 2 diabetes in order to set adequate preventive strategies.

ELIGIBILITY:
Inclusion Criteria:

* Women aged over 18years old
* Women with the criteria of GDM during pregnancy at 21-35 weeks of gestation (one situation):

  * After a 75g Oral Glucose Tolerance Test (OGTT - WHO criteria) with blood glucose (BG) values at T60≥180mg/dl and/or T120≥153mg/dl
  * An O. Sullivan test following a 100g oral glucose load with at least two pathological values (T60 ≥ 180mg/dl and/or T120 ≥ 155mg/dl and/or T180 ≥ 140mg/dl)
  * With a fasting BG value ≥92mg/dl
* Women with signed informed consent

Exclusion Criteria:

* Women aged less than 18years old
* Women with pregestational type 2 diabetes
* Women without signed informed consent
* Women who does not read and/or understand french language
* Women not affiliated to the health care system
* Women with recent infection (<1month) and/or on steroids or anti-inflammatory drugs.
* Women with chronic diseases
* Women with a disable state
* Women with normal glucose tolerance
* Women already incorporated in another clinical study that could interfere with the present study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2011-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Metabolic index value | 3 months after delivery (+/- 15 days)
  The primary objective relies on Receiver Operating Characteristic (ROC) curves of metabolic index values using peripheral markers during gestation : C-Reactive Protein ultrasensitive (CRPus), malonaldehyde (MDA) and adiponectin (index = (CRP + MDA)/adiponectin) to detect an abnormal glucose tolerance at 3 months (+/- 15 days) after delivery (M3) during a 75g oral glucose tolerance test (T0>110mg/dl and/or T120 >145mg/dl). The rationale for the index relies on lower adiponectin values high CRPus levels and MDA values during insulin resistance chronic inflammatory status and oxidative stress.

SECONDARY OUTCOMES:
Prevalence of abnormal glucose tolerance in women with GDM | 3 months (+/- 15 days) following delivery

OTHER OUTCOMES:
Prevalence of type 2 diabetes in women with GDM. | 18 months (+/- 2 months) after delivery
  Prevalence of women with fasting blood glucose levels > 126mg/dl at 18 months (+/- 2 months) after delivery.
Adiponectin level | 18 months (+/- 2 months) after delivery

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Hospices Civils de Lyon - Hôpital Femme-Mère-Enfant - Service de gynécologie obstétrique, Bron
  - CHU Clermont-Ferrand - Hôpital Gabriel Montpied - Service d'endocrinologie, Clermont-Ferrand
  - Centre Hospitalier de Givors - Hôpital de Montgelas - Service de médicine 8, Givors
  - CHU Grenoble - Clinique d'Endocrinologie Diabétologie Nutrition, Grenoble
  - Hospices Civils de Lyon - Groupement Hospitalier Sud - Service d'Endocrinologie, Diabète, Nutrition, Pierre-Bénite
  - CHU Saint Etienne - Hôpital Nord - Service d'endocrinologie, diabètes, nutrition, Saint-Etienne
  - Groupement Hospitalier des Portes du Sud - Service d'Endocrinologie Diabétologie Nutrition, Vénissieux

REFERENCES:
- [Result] Honnorat D, Disse E, Millot L, Mathiotte E, Claret M, Charrie A, Drai J, Garnier L, Maurice C, Durand E, Simon C, Dupuis O, Thivolet C. Are third-trimester adipokines associated with higher metabolic risk among women with gestational diabetes? Diabetes Metab. 2015 Nov;41(5):393-400. doi: 10.1016/j.diabet.2015.03.003. Epub 2015 Apr 15. PMID 25890778